CLINICAL TRIAL: NCT05243888
Title: A Randomised Controlled Trial Assessing the Efficacy of Strategies Involving Self-sampling to Reach Women Not Participating in Regular Cervical Cancer Screening
Brief Title: Efficacy of Strategies Involving Self-sampling to Reach Women Not Participating in Regular Cervical Cancer Screening
Acronym: CapU4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Regional de Coordination des Depistages des Cancer - Pays de la Loire (Other)
Collaborators: National Cancer Institute, France (Other Government); Sciensano (Other Government); University Hospital, Angers (Other Government); University of Angers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2021-A01660-41
Record Dates: First submitted 2022-01-26; First posted 2022-02-17 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Cancer Screening Test
Keywords: cervical cancer; screening coverage; cancer screening test; under-screened women; urinary self-sampling; vaginal self-sampling; randomised controlled trial; semi-structured interviews
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a randomised controlled trial with three arms: a control arm (conventional invitation letter) and two experimental arms (mailing of a urine or vaginal self-sampling kit).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control (No Intervention): The control arm corresponds to women receive a conventional invitation letter sent by post to the home address of eligible women recommending them to make an appointment to a doctor or a midwife for the collection of a cervical specimen.
- vaginal self-sampling (Experimental): eligible women receive at their home address a vaginal self-sampling kit in addition to the conventional invitation letter
  Interventions: Diagnostic Test: self-sampling
- urinary self-sampling (Experimental): eligible women receive at their home address a urine collection kit in addition to the conventional invitation letter
  Interventions: Diagnostic Test: self-sampling

INTERVENTIONS:
Diagnostic Test: self-sampling — eligible women receive at their home address a self-sampling kit in addition to the conventional invitation letter
  Arms: urinary self-sampling; vaginal self-sampling

SUMMARY:
The cervical cancer screening coverage remains moderate (60%) in France. The aim of the study is to evaluate the efficacy of two experimental invitation strategies (offer of urine or vaginal self-sampling kits) to reach under-screened populations and compare them with the current invitation strategy in rural departments (low medical density and low participation rate) in France.

The study is a randomised controlled trial with three arms: a control arm (conventional invitation letter) and two experimental arms (mailing of a urine or vaginal self-sampling kit). The target population includes women aged 30-65 years, who had no screening test recorded since more than four years and who did not respond to an invitation letter within twelve months before. The primary outcome measure is the participation rate in each arm.

A team of psychologists will also investigate attitudes and experiences by semi-structured/focus-group interviews with voluntary CapU4 participants and with health professionals.

CapU4 will identify effective strategies to reach women not responding to current screening invitations and will generate information about acceptance of self-sampling among women and health professionals.

DETAILED DESCRIPTION:
Research question: does the offer of self-sampling kits result in higher attendance to cervical cancer screening compared to sending invitation letters which recommend women to contact a health professional for taking a cervical specimen?

Systematic reviews indicate that Human Papillomavirus (HPV) testing on vaginal specimens taken by the woman her-self is as accurate to detect cervical precancer as HPV testing of cervical specimens collected by a clinician, under the condition that a validated polymerase chain reaction (PCR)-based HPV assay is used. Similar results are shown from recent studies where HPV testing was performed on first-void urine collected with an appropriate device and transport medium. A recent meta-analysis of randomised trials showed higher response rates when under-screened women receive a self-sampling kit at home compared to traditional invitation or reminder letters. However, the absolute participation rates are highly variable among studies. Whereas qualitative research indicates that women prefer collection of urine rather than a vaginal self-sample, no data are available that the offer of urine kits would result in higher participation among women who do not participate regularly in cervical cancer screening.

Objectives:

* To evaluate the effectiveness of two experimental invitation strategies (urine or vaginal self-sampling) to reach under-screened populations and compare them to the current invitation strategy in rural departments in France.
* To improve the response rate among women aged 30 to 65 years (not screened over a period longer than the recommended screening interval) who did not respond to a conventional prior invitation.

Trial design:

1:1:1 randomised population-based participation trial, with 2 experimental and 1 control arm, with in each arm a 1:1 sub-randomisation with subgroup A receiving a questionnaire and subgroup B receiving no questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 30 and 65 years
* living in the Departments of Mayenne, Vendée and Sarthe (Pays de la Loire, France)
* who have not carried out a screening test (cytology of smear or HPV test) following a letter sent 12 months previously (in 2020 or 2021).

Exclusion Criteria:

* recent cervical sampling (less than three years old)
* women younger than 30 or older than 65 years
* women who have had a hysterectomy
* women with ongoing follow-up for a cervical lesion
* women who are not members or beneficiaries of a social security system.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Rate of participation in each arm (%) | 6 months
  (number of responding / number of invited)

SECONDARY OUTCOMES:
Rate of participation (%) | 6 months
  (number of responding / number of invited). Contrast in participation between the 2 experimental arms
Rate of participation (%) with questionnaire or not | 6 months
  (number of responding / number of invited). Contrast in participation between women that received a questionnaire or not
Rate of screen test positivity (%) | 24 months
  Virological result. presence of high-risk HPV
Percentage of women screened positive with adherence to gynecological follow-up | 24 months
  gynecological follow-up (cytological results)
Impact of age on the participation (rate of participation %) | 6 months
  age
Impact of age on the adherence to gynecological follow-up (% of women) | 24 months
  age
Impact of reimbursement status on the participation (rate of participation %) | 6 months
  reimbursement status (benefit or not from supplementary universal health care coverage)
Impact of reimbursement status on the adherence to gynecological follow-up (% of women) | 24 months
  reimbursement status (benefit or not from supplementary universal health care coverage)
Impact of geographical area on the participation (rate of participation %) | 6 months
  geographical area (including the deprivation index corresponding with the statistical sector where the woman is domiciled)
Impact of geographical area on the adherence to gynecological follow-up (% of women) | 24 months
  geographical area (geographical area (including the deprivation index corresponding with the statistical sector where the woman is domiciled)
Obstacles and levers emerging from the speech of the women participating in the research (thematic analysis) | 24 months
  thematic analysis integrating a specific focus on the indicators identified in previous studies (e.g. lack of time, discomfort with regard to the location or bad experience encountered during another type of examination, etc.).
Obstacles and levers emerging from the speech of the women participating in the research (categorical analysis) | 24 months
  categorical analysis based on Linguistic Inquiry and Word count which allows, among other things, to automatically categorise positive or negative emotions related to themes for example associated with the disease or beliefs
Obstacles and levers emerging from the speech of the health professionals participating in the research (thematic analysis) | 24 months
  thematic analysis integrating a specific focus on the indicators identified in previous studies (e.g. lack of time, discomfort with regard to the location or bad experience encountered during another type of examination, etc.).
Obstacles and levers emerging from the speech of the health professionals participating in the research (categorical analysis) | 24 months
  categorical analysis based on Linguistic Inquiry and Word count which allows, among other things, to automatically categorise positive or negative emotions related to themes for example associated with the disease or beliefs

CONTACTS AND LOCATIONS:
Locations (1):
- CRCDC Pays de la Loire, Angers, France